CLINICAL TRIAL: NCT03203967
Title: Effect of Low-dose Epidural Morphine Combined With Single-injection Femoral Nerve Block on Postoperative Analgesia in Patients After Total Knee Arthroplasty
Brief Title: Epidural Morphine for Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017[1308]
Record Dates: First submitted 2017-05-30; First posted 2017-06-29 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Adult Patients; Total Knee Arthroplasty; Epidural Analgesia; Femoral Nerve Block; Analgesic Adverse Reaction
Keywords: Adults; Unilateral TKA; Single femoral nerve block; Low-dose epidural morphine; Effect of postoperative analgesia; Quality of life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural morphine (Experimental): 1. Epidural morphine (2 mg morphine in 5 ml normal saline) is administered through the epidural catheter at the end of surgery.
  2. Single femoral nerve block is performed with 20 ml of 0.5% ropivacaine under the guidance of ultrasonography and nerve stimulator after surgery.
  3. Intravenous morphine analgesia is provided with a patient-controlled analgesia pump which is established with 100 ml of 0.5 mg/mL morphine, programmed to deliver a 2 ml bolus with a lockout interval of 8-10 min and a background infusion of 0.5 mL/h.
  Interventions: Procedure: Epidural morphine; Procedure: Single femoral nerve block; Drug: Intravenous morphine analgesia
- Epidural placebo (Placebo Comparator): 1. Epidural placebo (5 ml normal saline) is administered through the epidural catheter at the end of surgery.
  2. Single femoral nerve block is performed with 20 ml of 0.5% ropivacaine under the guidance of ultrasonography and nerve stimulator after surgery.
  3. Intravenous morphine analgesia is provided with a patient-controlled analgesia pump which is established with 100 ml of 0.5 mg/mL morphine, programmed to deliver a 2 ml bolus with a lockout interval of 8-10 min and a background infusion of 0.5 mL/h.
  Interventions: Procedure: Epidural placebo; Procedure: Single femoral nerve block; Drug: Intravenous morphine analgesia

INTERVENTIONS:
Procedure: Epidural morphine — 2 mg of morphine (0.4 mg/ml morphine in 5 ml normal saline) is administered through the epidural catheter at the end of surgery.
  Arms: Epidural morphine
Procedure: Epidural placebo — 5 ml normal saline is administered through the epidural catheter at the end of surgery.
  Arms: Epidural placebo
Procedure: Single femoral nerve block — Single femoral nerve block is performed with 20 ml 0.5% ropivacaine under the guidance of ultrasonography and nerve stimulator after surgery.
Drug: Intravenous morphine analgesia — Intravenous morphine analgesia is provided with a patient-controlled analgesia pump which is established with 100 ml of 0.5 mg/ml morphine, programmed to deliver a 2 ml bolus with a lockout interval of 8-10 min and a background infusion of 0.5 ml/h.

SUMMARY:
Single femoral nerve blockade combined with patient-controlled intravenous analgesia are used for postoperative analgesia for patients after TKA in the hospital of the investigators. Although this method provides acceptable analgesia, the incidence of opioid-associated side effects is relatively high. Low-dose epidural morphine is commonly used in postoperative analgesia after cesarean section, and the effect of single dose morphine lasts more than 20 hours, with low incidences of itching, nausea, vomiting, and respiratory depression. The investigators hypothesize that, for patients undergoing TKA, the addition of low-dose epidural morphine to single femoral nerve block and intravenous opioids can improve the postoperative analgesia, reduce the consumption of intravenous opioids and decrease opioid-associated side effects.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is an important therapy for patients with serious knee osteoarthritis in order to improve quality of life and relieve pain. But a large number of patients who undergo this surgery experience moderate to severe postoperative pain. Previously, the investigators used single femoral nerve blockade combined with patient-controlled intravenous analgesia for postoperative analgesia for patients after TKA. Although this method provides acceptable analgesia, the incidence of opioid-associated side effects is relatively high. Low-dose epidural morphine is commonly used in postoperative analgesia after cesarean section, and the effect of single dose morphine lasts more than 20 hours, with low incidences of itching, nausea, vomiting, and respiratory depression. The investigators hypothesize that, for patients undergoing TKA, the addition of low-dose epidural morphine to single femoral nerve block and intravenous opioids can improve the postoperative analgesia, reduce the consumption of intravenous opioids and decrease opioid-associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age of 18 years or older);
* American Society of Anesthesiologists classification I-III;
* Scheduled to undergo unilateral TKA under combined spinal and epidural anesthesia.

Exclusion Criteria:

* Age higher than 90 years old;
* Presence of any contraindication to neuraxial block or peripheral nerve block;
* Continuous use of opioid analgesics during the last month;
* Unable to understand Numeric Rating Scale for pain evaluation or existence of language barrier;
* Severe renal insufficiency (requirement of renal replacement therapy);
* History of asthma;
* Recruited in another clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Percent of patients with moderate to severe pain (Numeric Rating Scale pain score of 4 or higher) | Until 48 hours after surgery.
  Pain severity is evaluated with Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) both at rest and with movement.

SECONDARY OUTCOMES:
NRS pain scores (at rest and with movement) at various timepoints after surgery | At 6, 12, 24, 36 and 48 hours after surgery.
  Pain severity is evaluated with Numeric Rating Scale (NRS, an 11-point scale where 0 = no pain and 10 = the worst pain) both at rest and with movement.
Cumulative morphine consumption | Until 48 hours after surgery.
  Cumulative morphine consumption during 48 hours after surgery.
Recovery of motor function of the lower limb from blockade | At the end of the surgery and at 0.5, 6, 12, 24, 36, 48 hours after surgery.
  Modified Bromage scale (0 = no blockade: extended limb lift off the bed; 1 = flexion/extension at knee and ankle joint; 2 = no flexion/extension at knee or ankle joint; 3 = complete blockade).
Time to begin functional exercise and ground walking | During hospital stay, up to 1 week after surgery.
  Time to begin functional exercise and ground walking
Patient's satisfaction with analgesia | At 48 hours after surgery.
  Evaluated in 5 scale, i.e., very satisfactory, satisfactory, neither satisfactory nor unsatisfactory, unsatisfactory, and very satisfactory.
Length of stay in hospital after surgery | Until hospital discharge up to 30 days after surgery.
  Length of stay in hospital after surgery
Incidence of postoperative complication | Until 30 days after surgery.
  Incidence of postoperative complication within 30 days after surgery.
The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index | At 30 days after surgery.
  Evaluated with the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index.
Quality of life (SF-12) at 30 days after surgery | At 30 days after surgery.
  Evaluated with Short-Form Health Survey-12 (SF-12) at 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamplot JD, Wagner ER, Manning DW. Multimodal pain management in total knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Feb;29(2):329-34. doi: 10.1016/j.arth.2013.06.005. Epub 2013 Jul 11. PMID 23850410
- [Background] Dong CC, Dong SL, He FC. Comparison of Adductor Canal Block and Femoral Nerve Block for Postoperative Pain in Total Knee Arthroplasty: A Systematic Review and Meta-analysis. Medicine (Baltimore). 2016 Mar;95(12):e2983. doi: 10.1097/MD.0000000000002983. PMID 27015172
- [Background] Pulos N, Sheth N. Perioperative pain management following total joint arthroplasty. Ann Orthop Rheumatol. 2014;2(3):1029.Google Scholar
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Wang H, Boctor B, Verner J. The effect of single-injection femoral nerve block on rehabilitation and length of hospital stay after total knee replacement. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):139-44. doi: 10.1053/rapm.2002.29253. PMID 11915059
- [Background] Bonica J. Postoperative pain. In: Bonica J, editor. The Management of Pain. 2nd ed. Philadelphia: Lea & Febiger; 1990. p. 461-80.
- [Background] Pang WW, Hsu TC, Tung CC, Hung CP, Chang DP, Huang MH. Is total knee replacement more painful than total hip replacement? Acta Anaesthesiol Sin. 2000 Sep;38(3):143-8. PMID 11125689
- [Background] Chughtai M, Jauregui JJ, Mistry JB, Elmallah RK, Diedrich AM, Bonutti PM, Delanois R, Mont MA. What Influences How Patients Rate Their Hospital After Total Knee Arthroplasty? Surg Technol Int. 2016 Apr;28:261-5. PMID 27042784
- [Background] Lavie LG, Fox MP, Dasa V. Overview of Total Knee Arthroplasty and Modern Pain Control Strategies. Curr Pain Headache Rep. 2016 Nov;20(11):59. doi: 10.1007/s11916-016-0592-6. PMID 27655139
- [Background] Seet E, Leong WL, Yeo AS, Fook-Chong S. Effectiveness of 3-in-1 continuous femoral block of differing concentrations compared to patient controlled intravenous morphine for post total knee arthroplasty analgesia and knee rehabilitation. Anaesth Intensive Care. 2006 Feb;34(1):25-30. doi: 10.1177/0310057X0603400110. PMID 16494145
- [Background] Tierney E, Lewis G, Hurtig JB, Johnson D. Femoral nerve block with bupivacaine 0.25 per cent for postoperative analgesia after open knee surgery. Can J Anaesth. 1987 Sep;34(5):455-8. doi: 10.1007/BF03014348. PMID 3664912
- [Background] Weber A, Fournier R, Van Gessel E, Gamulin Z. Sciatic nerve block and the improvement of femoral nerve block analgesia after total knee replacement. Eur J Anaesthesiol. 2002 Nov;19(11):834-6. doi: 10.1017/s0265021502221353. No abstract available. PMID 12442936
- [Background] Mansour NY, Bennetts FE. An observational study of combined continuous lumbar plexus and single-shot sciatic nerve blocks for post-knee surgery analgesia. Reg Anesth. 1996 Jul-Aug;21(4):287-91. PMID 8837184
- [Background] Sundarathiti P, Ruananukul N, Channum T, Kitkunasathean C, Mantay A, Thammasakulsiri J, Sodsee W. A comparison of continuous femoral nerve block (CFNB) and continuous epidural infusion (CEI) in postoperative analgesia and knee rehabilitation after total knee arthroplasty (TKA). J Med Assoc Thai. 2009 Mar;92(3):328-34. PMID 19301724
- [Background] Popping DM, Zahn PK, Van Aken HK, Dasch B, Boche R, Pogatzki-Zahn EM. Effectiveness and safety of postoperative pain management: a survey of 18 925 consecutive patients between 1998 and 2006 (2nd revision): a database analysis of prospectively raised data. Br J Anaesth. 2008 Dec;101(6):832-40. doi: 10.1093/bja/aen300. Epub 2008 Oct 22. PMID 18945716
- [Background] Duarte VM, Fallis WM, Slonowsky D, Kwarteng K, Yeung CK. Effectiveness of femoral nerve blockade for pain control after total knee arthroplasty. J Perianesth Nurs. 2006 Oct;21(5):311-6. doi: 10.1016/j.jopan.2006.05.011. PMID 17027440
- [Background] Salinas FV, Liu SS, Mulroy MF. The effect of single-injection femoral nerve block versus continuous femoral nerve block after total knee arthroplasty on hospital length of stay and long-term functional recovery within an established clinical pathway. Anesth Analg. 2006 Apr;102(4):1234-9. doi: 10.1213/01.ane.0000198675.20279.81. PMID 16551930
- [Background] Soto Mesa D, Del Valle Ruiz V, Fayad Fayad M, Cosio Carreno F, Blanco Rodriguez I, Gonzalez Castano R, Bermejo Alvarez MA. [Control of postoperative pain in knee arthroplasty: single dose femoral nerve block versus continuous femoral block]. Rev Esp Anestesiol Reanim. 2012 Apr;59(4):204-9. doi: 10.1016/j.redar.2012.02.013. Epub 2012 Apr 30. Spanish. PMID 22551482
- [Background] Singh SI, Rehou S, Marmai KL, Jones APM. The efficacy of 2 doses of epidural morphine for postcesarean delivery analgesia: a randomized noninferiority trial. Anesth Analg. 2013 Sep;117(3):677-685. doi: 10.1213/ANE.0b013e31829cfd21. Epub 2013 Aug 6. PMID 23921652
- [Background] Marroquin B, Feng C, Balofsky A, Edwards K, Iqbal A, Kanel J, Jackson M, Newton M, Rothstein D, Wong E, Wissler R. Neuraxial opioids for post-cesarean delivery analgesia: can hydromorphone replace morphine? A retrospective study. Int J Obstet Anesth. 2017 May;30:16-22. doi: 10.1016/j.ijoa.2016.12.008. Epub 2016 Dec 30. PMID 28185794
- [Background] Sundarathiti P, Thammasakulsiri J, Supboon S, Sakdanuwatwong S, Piangjai M. Comparison of continuous femoral nerve block (CFNB/SA) and continuous femoral nerve block with mini-dose spinal morphine (CFNB/SAMO) for postoperative analgesia after total knee arthroplasty (TKA): a randomized controlled study. BMC Anesthesiol. 2016 Jul 16;16(1):38. doi: 10.1186/s12871-016-0205-2. PMID 27422406
- [Derived] Meng ZT, Cui F, Li XY, Wang DX. Epidural morphine improves postoperative analgesia in patients after total knee arthroplasty: A randomized controlled trial. PLoS One. 2019 Jul 1;14(7):e0219116. doi: 10.1371/journal.pone.0219116. eCollection 2019. PMID 31260468